CLINICAL TRIAL: NCT02318862
Title: Assessment of Esophageal Epithelium Integrity With Mucosal Impedance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Michael Vaezi, Principal Investigator, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 130084
Record Dates: First submitted 2013-09-04; First posted 2014-12-17 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Gastroesophageal Reflux Disease (GERD); Non-erosive Reflux Disease (NERD)
Keywords: reflux; GERD; EGD; pH testing
MeSH Terms: conditions — Gastroesophageal Reflux; Non-Erosive Reflux Disease | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GERD (Other): Those who have abnormal pH and abnormal esophageal mucosa and those who have abnormal pH and normal esophageal mucosa and are scheduled for standard of care esophagogastroduodenoscopy (EGD) with mucosal impedance testing
  Interventions: Procedure: Standard of Care esophagogastroduodenoscopy (EGD) with mucosal impedance testing
- non-GERD (Other): Those who have normal pH and normal esophageal mucosa and are scheduled for standard of care esophagogastroduodenoscopy (EGD) with mucosal impedance testing
  Interventions: Procedure: Standard of Care esophagogastroduodenoscopy (EGD) with mucosal impedance testing

INTERVENTIONS:
Procedure: Standard of Care esophagogastroduodenoscopy (EGD) with mucosal impedance testing

SUMMARY:
Gastroesophageal reflux disease (GERD) is a common condition affecting more than 100 million adults in the U.S., and it significantly impacts patients' quality of life while imposing billions of dollars of direct and indirect costs each year upon our healthcare system. Current diagnostic tests for GERD are highly invasive and medically inadequate, and the goal of this project is to develop a novel, minimally invasive Mucosal Impedance technique for more accurate detection of GERD while reducing costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing standard of care EGD with 48-hr pH testing by BRAVO
* Previous diagnosis of reflux
* At least 18 years of age

Exclusion Criteria:

* Those less than 18 years of age
* Unable to give informed consent
* Use of acid suppressive therapy within the last 10 days
* Known history of Barrett's esophagus, gastric surgery, alcoholism, or significant motility condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Measurement of lower esophageal impedance using mucosal impedance catheter | During standard of care EGD
  Mucosal impedance is obtained during routine care EGD and readings are compared to 48-hour Bravo capsule results. Mucosal impedance only takes one minute to perform during endoscopy.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Vaezi, MD, PhD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No